CLINICAL TRIAL: NCT02557685
Title: Alterations in Gut Microbiota and Metabolism Following FMT for Recurrent C. Difficile Infection
Brief Title: Gut Microbiota Changes After Fecal Microbiota Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Colleen Kelly, Medical Doctor, The Miriam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16216
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Translantation (No Intervention): After completing at least 10 days course of antibiotic treatment for C. difficile infection, subjects will receive Fecal Microbiota transplantation with a 300 mL fecal suspension delivered via sigmoidoscopy.
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal Microbiota Translantation involves administering fecal material from a healthy donor to a sick patient, with relapsing C-difficile infection, to restore missing components of normal intestinal flora. Subjects will receive Fecal Microbiota Translantation via sigmoidoscopy.
  Other Names: FMT, stool transplant

SUMMARY:
This study aims to document early changes in the distal gut microbiota (both fecal and mucosa-associated) post FMT. Furthermore, whole blood and urine samples will facilitate collaborative immunologic and metabolomic analyses.

This will be an open label clinical trial of FMT to prevent further recurrence in patients who have suffered at least a third episode of Clostridium difficile infection (CDI) and who have previously been treated with oral vancomycin.

DETAILED DESCRIPTION:
The exact mechanism by which FMT is effective is presently unknown. A recent study of 14 patients with recurrent CDI treated with FMT35 showed decreased diversity pre-FMT with gut microbiota becoming more diverse and similar to donors post-FMT. This group showed significant changes in 3 taxonomic orders but no single organism or species was universally associated with success. Weingarden et al. showed that FMT restored normal bile acid composition in patients with recurrent CDI36, suggesting that correction of bile acid metabolism is likely a major mechanism by which FMT results in a cure and prevents recurrence of CDI. Understanding mechanisms of FMT more completely may enable development of synthetic microbiota-based therapeutics which would be a safe and effective alternative to traditional FMT. We hypothesize that early changes in distal gut microbiota post-FMT may help identify key species associated with efficacy. Furthermore, we believe there are measurable metabolic and immunologic effects which may also be beneficial after FMT. This study aims to document early changes in the distal gut microbiota (both fecal and mucosa-associated) post FMT. Furthermore, whole blood and urine samples will facilitate collaborative immunologic and metabolomic analyses.

This will be an open label clinical trial of FMT to prevent further recurrence in patients who have suffered at least a third episode of Clostridium difficile infection (CDI) and who have previously been treated with oral vancomycin. Subjects will consist of 6 adult outpatients referred after 3 (or more) episodes of CDI. Subjects, who will have been treated with at least a 10 day course of anti-CDI therapy (metronidazole, vancomycin or fidaxomicin) for the most recent acute infection, will then receive FMT with donor stool administered at the time of sigmoidoscopy. After the procedure, subjects will be followed for 8 weeks for C. difficile recurrence. Subjects who relapse during that period will be offered a repeat FMT using donor stool. We plan to collect baseline and post-FMT stool samples for microbiome analyses as well samples of urine and blood for metabolomic and immunologic studies. Subjects will be contacted at 24 weeks to assess long term safety outcomes

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (age ≥18 and ≤90) referred to Dr. Kelly after suffering a third (or further) documented episode CDI and 2) who have failed to maintain CDI cure after standard therapy.

  * Previous treatment with at least one course of tapered/pulse dose vancomycin as per SHEA-IDSA C difficile treatment guidelines or
  * Inability to taper or stop anti-CDI therapy without developing diarrhea requiring anti-infective therapy

Exclusion Criteria:

* • Patients who are pregnant

  * Patients who are nursing
  * Patients who are incarcerated
  * Patients with cognitive impairment or severe neuropsychiatric co morbidities who are incapable of giving their own informed consent
  * Patients who are immunocompromised specifically:

    * HIV infection (any CD4 count)
    * AIDS-defining diagnosis or CD4<200/mm3
    * Inherited/primary immune disorders
    * Immunodeficient or Immunosuppressed due to medical condition/medication:
    * Current or recent (<3 most) treatment with anti-neoplastic agent
    * Current or recent (<3 mos) treatment with any immunosuppressant medications (including but not limited to monoclonal antibodies to B and T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil). Subjects who are otherwise immunocompetent and have discontinued any immunosuppressant medications 3 or more months prior to enrollment may be eligible to enroll.
  * Patients with a history of severe (anaphylactic) food allergy
  * Patients who have previously undergone FMT
  * Patients who are unwilling or unable to undergo sigmoidoscopy
  * Patients with untreated, in-situ colorectal cancer
  * Patients with a history of inflammatory bowel disease (ulcerative colitis, Crohn's disease or microscopic colitis) or diarrhea-predominant irritable bowel syndrome
  * Unable to comply with protocol requirements
  * Patients who are American Society of Anesthesiologists (ASA) Physical Status classification IV and V
  * Patients with acute illness or fever on the day of planned FMT will be excluded (not undergo randomization or treatment with FMT) with the option of including that subject at a future date.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Clinical cure | 8 weeks

SECONDARY OUTCOMES:
Clinical failure | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelly, MD, Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States